CLINICAL TRIAL: NCT03075137
Title: Effect of External Counter Pulsation on IschemicStroke (ECP-STROKE)
Brief Title: Effect of External Counter Pulsation on Ischemic Stroke
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Chinese University of Hong Kong (Other); Second Affiliated Hospital of Xi'an Jiaotong University (Other); Second Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Guifu Wu, Eighth Affiliated Hospital, Sun Yat-Sen University, Eighth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SYSU8002
Record Dates: First submitted 2017-02-28; First posted 2017-03-09 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-12

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; external counter pulsation; mRS
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- External Counter Pulsation (ECP) group (Experimental): A standard ECP protocol involves 35 one-hour sessions (once per day, 5 days a week) and continuous for 7 weeks. ECP consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading.
  Interventions: Device: External counter pulsation (ECP)
- Control group (No Intervention): Guideline-driven standard medical treatment

INTERVENTIONS:
Device: External counter pulsation (ECP) — standard ECP protocol involves 35 one-hour sessions (once per day, 5 days a week) and continuous for 7 weeks. ECP consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading.
  Arms: External Counter Pulsation (ECP) group

SUMMARY:
Stroke is a prevalent atherosclerosis vascular disease with high mortality, external counter pulsation (ECP) is an approved noninvasive therapy for angina, congestive heart failure, myocardial infarction, and cardiogenic shock that augments blood flow to cardiac and systemic circuits, which improves the flow volume in the carotid. Though ECP is Ⅱa recommendation for stroke management, no multi-center control clinical study has been reported for prognosis of stroke. The aim of this study is to evaluate the effect of ECP on stoke. To address this assumption, investigators enroll subjects with ischemic stroke and randomized into control or ECP group, the ECP intervention will be carried out with a standard protocol which involves 35 one-hour sessions (5 days a week) for continuous 7 weeks. The primary endpoint is mRS score in 3 months, secondary endpoints include NIHSS, BI and MMSE score, recurrence of stroke in 3 months, glycolipid metabolism, transcranial doppler (TCD) flow velocities and endothelial function.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of mortality worldwide, accounting for 17.5 million deaths per year; 6.7 million of these deaths are related to stroke. Over 80% of strokes are classified as ischemic. External counter pulsation (ECP) is a non-invasive method which consists of three sets of pneumatic cuffs attached to each of the patient's legs at the calf and lower and upper thigh. The inflation of the cuffs is triggered by a computer, and timing of the inflation is based on the R wave of the electrocardiogram. The ECP therapist adjusts the inflation and deflation timing to provide optimal blood movement per a finger plethysmogram waveform reading. This produces a retrograde flow of blood in the aorta resulting in a diastolic augmentation of blood flow and also an increase in venous return, which leads to an improved carotid perfusion pressure. Cumulative evidences demonstrate that ECP can augment peak diastolic and mean middle cerebral artery flow velocities, accelerate rehabilitation after stroke, however, no multi-center study on the effect of ECP on the prognosis of stroke has been reported. Thus, this study is designed to enroll 380 subjects with ischemic stroke after evaluation of glycolipid metabolism, heart function, transcranial doppler (TCD) flow velocities, endothelial function, NIHSS, BI and MMSE score, they will be randomized into ECP intervention or control group. All subjects receive Guideline-driven standard medical treatment, ECP will be carried out with a standard protocol which involves 35 one-hour sessions (5 days a week) for continuous 7 weeks. Up to the end of ECP intervention, mRS of subjects will be follow up to 3 months, meanwhile, items as above will be retested for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ischemic stroke
* Exclusion cerebral hemorrhage after CT scan
* NIH Stroke Scale (NIHSS)≥4
* Modified Rankin Scale (mRS) 0-1
* Signed informed consent

Exclusion Criteria:

* Obvious aortic insufficiency;
* Aortic aneurysm or aortic dissection;
* Coronary fistula or severe coronary aneurysm;
* Not controlled bleeding disease with INR>2.0 ;
* Symptomatic Congestive heart failure
* Valvular heart disease, congenital heart diseases, cardiomyopathies
* Cerebral hemorrhage within six months;
* Uncontrolled hypertension, defined as SBP≥180mmHg or DBP≥110mmHg;
* Lower limb infection;
* Deep venous thrombosis;
* Progressive malignancies or diseases with poor prognosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2018-06-10 (Estimated); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale （mRS） score | Change from Baseline at 3 months
  3-month mRS score after stroke

SECONDARY OUTCOMES:
NIH Stroke Scale (NIHSS) score | Change from Baseline at 3 months
  3-month NIHSS score after stroke
Barthel Index (BI) | Change from Baseline at 3 months
  3-month BI after stroke
mini-mental state examination (MMSE) Score | Change from Baseline at 3 months
  3-month MMSE after stroke
Ischemic area of Cerebral CT image | Change from Baseline at 3 months
  Ischemic area of 3-month Cerebral CT image
Transcranial doppler (TCD) flow velocities | Change from Baseline at 3 months
  transcranial doppler (TCD) flow velocities

CONTACTS AND LOCATIONS:
Overall Officials: Guifu Wu, PhD, Study Chair — Eighth Affiliated Hospital, Sun Yat-sen University
Locations (3):
- China (3):
  - Shenzhen Research Institute, The Chinese University Hong Kong, Shenzhen, Guangdong
  - The Second Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: Undecided